CLINICAL TRIAL: NCT06928545
Title: Post-Market Assessment of the Incidence and Severity of Internal Hernia and Bowel Obstruction at One Year Following Use of the MagDI System to Create Side-to-Side Duodeno-Ileal Magnetic Compression Anastomoses (MagDI US Registry)
Brief Title: MagDI U.S. Registry
Status: Recruiting | Type: Observational
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GTM-007
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Anastomosis, Surgical; Internal Hernia; Bowel Obstruction
Keywords: GT Metabolic; MagDI System; Magnetic Anastomosis
MeSH Terms: conditions — Internal Hernia; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MagDI System: Participants who underwent the MagDI System procedure and consented to participate in the Registry
  Interventions: Device: Side-to-side duodenal-ileal anastomosis

INTERVENTIONS:
Device: Side-to-side duodenal-ileal anastomosis — Side-to-side duodenal-ileal anastomosis formed by magnetic compression using the GT Metabolic MagDI System.

SUMMARY:
Assess the incidence and severity of internal hernia and bowel obstruction at one year in a U.S. population following use of the MagDI System to create side-to-side duodeno-ileal anastomoses.

DETAILED DESCRIPTION:
Small bowel obstruction (SBO) following various abdominal and pelvic surgeries (0.4% - 13.9% at 5 years post-surgery) across obese and non-obese patients has been well studied in the scientific literature and found to be primarily due to intraperitoneal adhesions, with surgical technique (open surgery versus laparoscopic) cited as a key risk factor as reported in a retrospective population-based registry in Sweden (n=108,141). SBO incidence was reported as 3.2% for those undergoing bariatric surgery (n=1,896).

Given the MagDI System premarket clinical study (GTM-001) was conducted outside the U.S., FDA requires one post-market surveillance study to assess and characterize the incidence and severity of internal hernia and bowel obstruction in the U.S. intended use population treated with MagDI System. This study will be conducted through an observational patient registry and compare registry data to the premarket MagDI System clinical study data (GTM-001) and scientific literature. This post-market Registry Study was also a condition of the MagDI System FDA 510(k) clearances K242086 and K243359.

ELIGIBILITY:
Inclusion Criteria:

1. >21 years of age, at the time of informed consent.
2. Body Mass Index (BMI) between 30-50 kg/m2.
3. Indicated for a side-to-side duodeno-ileal anastomosis and is treated with the MagDI System at a U.S. registry center.
4. Participant has been informed of the nature of the registry.

Exclusion Criteria:

1. Participant does not provide informed consent to be enrolled and followed in the registry.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients in the U.S. who undergo a side-to-side duodeno-ileal anastomosis with the MagDI System.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Internal Hernia and Bowel Obstructions | From date of study index procedure through 360 days.
  To assess and characterize incidence and severity of internal hernia and bowel obstruction at one year in U.S. patients treated with the MagDI System compared with the pre-market study (GTM-001) and scientific literature.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Ventura Advanced Surgical Associates, Ventura, California
  - Baptist Healthcare System, Inc., Louisville, Kentucky
  - Ochsner Clinic Foundation, Lafayette, Louisiana
  - Bariatric Specialists of the Carolinas, Cary, North Carolina

IPD SHARING:
Plan to Share IPD: No